CLINICAL TRIAL: NCT04267588
Title: Using Technology to Track Pain and Pain-related Outcomes
Status: Recruiting | Type: Observational
Sponsor: Johns Hopkins University (Other)
Collaborators: PainCare, LLC (Unknown)
Responsible Party: Sponsor
Other Study IDs: IRB00196831
Record Dates: First submitted 2020-02-11; First posted 2020-02-13 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Pain, Chronic
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Navio App: The investigators propose to collect self-report and passively collected biological data and evaluate participants' relation to clinical and laboratory pain as well as patients' willingness to use and level of comfort with the mobile pain management digital platform and wearable biosensors. Eligible participants will be consented, given two biosensors (i.e., Apple Watch Series 1 with KardiaBand; Spire), a sleep monitoring device (actigraph watch), and a mobile app enabled smartphone, then trained on how to use the app (and device if appropriate) and biosensors. Participants will keep medications constant and not have any new pain treatment procedures over the course of the study period and 2 weeks prior to starting the study.
  Interventions: Other: Navio Mobile App

INTERVENTIONS:
Other: Navio Mobile App — Participants will use the Navio Mobile App to track participants' pain and pain treatment

SUMMARY:
Persistent pain is a public health epidemic. The current protocol seeks to develop technology to aid patients' tracking of patients' pain, medications and pain-related variables. The investigators seek to talk with patients in co-investigator's clinic to solicit feedback, as well as pilot test the technology with pain patients.

DETAILED DESCRIPTION:
Chronic pain affects over 100 million Americans, costs the US over $630 billion annually, and reduces quality of life. It is among the most clinically challenging and financially burdensome conditions facing clinicians and healthcare organizations. Sleep disturbance is common in chronic pain conditions with some studies reporting a prevalence as high as 70%-88%. Psychiatric disorders, including substance abuse and mood disorders are prevalent in chronic pain and are associated with impairment and decreased quality of life. Sleep is increasingly recognized as a critical regulator of mental health. Taken together, epidemiological, cross-sectional, and prospective studies support the hypothesis that insomnia, chronic pain, and depression are mutually interacting, each increasing the risk for the emergence and/or exacerbation of the other. The gold standard of chronic pain management is multidisciplinary pain treatment (MPT), but patients rarely receive MPT secondary to limited access and a severe shortage of pain management specialists. Thus, there is an urgent need for empirically supported, cost-effective multidisciplinary pain self-management options that are accessible to patients and trusted by primary and tertiary care providers. To address this problem, the investigators' group in collaboration with the Johns Hopkins Technology Innovation Center (TIC) has developed a mobile chronic pain, medication and symptom tracking digital technology platform designed to eventually support multidisciplinary pain treatment by enhancing patient-provider communication and delivering comprehensive, personalized, interactive evidence-based pain management strategies. The investigators' App (version 1.3) is currently able to collect self-report data (i.e., pain; sleep; mood; catastrophizing; stress; pain flares) and continuous, passively collected wearable biosensor data (i.e., heart rate; breathing; sleep; heart rate variability/stress). The investigators propose a prospective, observational proof of concept study to demonstrate feasibility and adherence while establishing the psychometric properties of a mobile pain App and to compare these data with passively collected physiological data and laboratory indices of pain in patients with chronic low back pain (CLBP).

ELIGIBILITY:
Inclusion Criteria:

* ≥ 21 years of age
* Pain duration > 3 months
* Average pain level of >3 out of 10 (0=no pain; 10=worst pain imaginable)
* English fluency
* Are not scheduled to undergo any medical procedures during the course of the study
* Have a physician-confirmed medical diagnosis associated with chronic pain
* Are willing to comply with the study protocol and give written informed consent. Patients taking non-narcotic analgesics must be on a stable dose one month prior to participation.

Exclusion Criteria:

* Delirium, dementia, or cognitive impairment (i.e., Mini Mental State Exam score <24)
* Unstable major psychiatric disorder or history of schizophrenia
* Beck Depression Inventory score >30 or report of suicidal ideation
* Active substance abuse;
* Refusal to provide access to relevant medical record information.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic low back pain (CLBP).
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-08-10 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Patterns of self-reported clinical Pain | Up to 2 weeks
  Patients will complete twice-daily, electronic (i.e. via mobile app) numerical pain rating scales through Navio App.
Patterns of Pain Catastrophizing | Up to 2 weeks
  Patients will complete twice-daily, electronic (i.e. via mobile app) pain catastrophizing questions through Navio App.
Patterns of Positive Mood | Up to 2 weeks
  Patients will complete twice-daily, electronic (i.e. via mobile app) positive mood questions through Navio App.
Patterns of Negative Mood | Up to 2 weeks
  Patients will complete twice-daily, electronic (i.e. via mobile app) negative mood questions through Navio App.

SECONDARY OUTCOMES:
Patient Adherence as assessed by completion of questionnaire on the app | Up to 2 weeks
  Daily and weekly patterns of electronic (i.e. mobile app) questionnaire completion will be assessed to determine compliance with the use of the app.

CONTACTS AND LOCATIONS:
Overall Officials: Luis F Buenaver, Ph. D, Principal Investigator — Johns Hopkins University
Locations (1):
- Behavioral Medicine Research Lab, Baltimore, Maryland, United States